CLINICAL TRIAL: NCT04655040
Title: A PHASE 1, 2-PERIOD, FIXED-SEQUENCE, MULTIPLE-DOSE, OPEN-LABEL STUDY TO ESTIMATE THE EFFECTS OF RITLECITINIB (PF-06651600) ON THE PHARMACOKINETICS OF A SINGLE DOSE OF CAFFEINE IN HEALTHY PARTICIPANTS
Brief Title: Estimation of the Effect of Multiple Dose Ritlecitinib (PF-06651600) on the Pharmacokinetics of a Single Dose of Caffeine in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B7981054
Record Dates: First submitted 2020-12-03; First posted 2020-12-04 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Caffeine; PF-06651600

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Caffeine and Ritlecitinib (Experimental): In Period 1 Day 1, participants will be dosed with a single oral administration of caffeine 100 milligram (mg) tablet.
  In Period 2 Day 1 to Day 7, participants will be dosed with a single oral administration of ritlecitinib 200 milligram (mg) tablet. On Day 8, participants will be dosed with caffeine 100 milligram (mg) tablet within 5 minutes after administration of a 200 milligram (mg) dose of ritlecitinib on the morning of Day 8. Dosing with oral 200 milligram (mg) ritlecitinib QD will continue until Day 9.
  Interventions: Drug: Caffeine; Other: Ritlecitinib

INTERVENTIONS:
Drug: Caffeine — 100milligram (mg) tablet taken orally in period 1 and period 2
Other: Ritlecitinib — 200 milligrams (mg) taken orally once a day(QD) for 8 days
  Other Names: PF-06651600

SUMMARY:
This will be a Phase 1, 2 period, fixed sequence, multiple-dose, open-label study of the effect of ritlecitinib on caffeine PK in healthy participants. Approximately 12 healthy male and/or female participants will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

-Male and female participants must be 18 to 55 years of age, inclusive, at the time of signing the ICD.

-BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb). -

* Male and female participants who are healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and 12-lead ECG.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, dermatological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* History of febrile illness within 5 days prior to the first dose of investigational product.
* History of any lymphoproliferative disorder such as EBV related lymphoproliferative disorder, history of lymphoma, history of leukemia, or signs or symptoms suggestive of current lymphatic or lymphoid disease.
* Known presence or a history of malignancy other than a successfully treated or excised non metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Participants who, according to the information provided on Drugs.com, would be at increased safety risk if dosed with caffeine.
* History of hypersensitivity to caffeine.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time profile from time 0 extrapolated to infinity (AUCinf) of caffeine | Day1 and Day8: Hour 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24. Day 8: Hour 36 and 48

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events | Baseline through Day 28
Incidence of clinically significant abnormalities in vital signs | Baseline through Day 11
Incidence of clinically significant abnormalities in clinical laboratory values | Baseline through Day 11

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981054